CLINICAL TRIAL: NCT05795335
Title: Survival Outcomes, Adverse Events and Predictive Biomarkers for CDK4/6 Inhibitors in Patients With Hormone Receptor-positive Advanced Breast Cancer, an Ambispective Single-center Cohort Study
Brief Title: CDK4/6 Inhibitors in Patients With Hormone Receptor-positive Advanced Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Lu, Jinsong Lu, Chief of Breast Surgery Department, RenJi Hospital, RenJi Hospital
Other Study IDs: KY2022-097-B
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: Locoregionally Recurrent; Metastatic; CDK4/6 Inhibitors
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients have received or plan to receive CDK4/6 inhibitors for advanced disease.
  Interventions: Drug: CDK4/6 inhibitor

INTERVENTIONS:
Drug: CDK4/6 inhibitor — CDK4/6 inhibitors

SUMMARY:
This is an ambispective, single-center study to evaluate the survival outcomes, adverse events and predictive biomarkers for CDK4/6 inhibitors in patients with hormone receptor-positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and older
* Confirmed diagnosis of hormone receptor-positive breast cancer.
* Subjects with locoregionally recurrent or metastatic disease not amenable to curative therapy.
* Subjects have received or plan to receive CDK4/6 inhibitors for advanced disease.
* ECOG 0-2
* Adequate organ function

Exclusion Criteria:

* Subjects disable to swallow pills.
* History of immunodeficiency disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hormone receptor-positive breast cancer patients who have received or plan to receive CDK4/6 inhibitors for advanced disease.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of starting CDK4/6 inhibitor to the date of first documentation of progression or death (up to approximately 2.5 years)
  PFS is defined as the time from the date of starting CDK4/6 inhibitor to the date of objective tumor progression as per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) or death from any cause in the absence of documented PD, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | From the date of starting CDK4/6 inhibitor until death from any cause up to 3 years
  Overall survival is defined as the time from starting CDK4/6 inhibitor to death from any cause.
Adverse events | From the date of starting CDK4/6 inhibitor to the end of the treatment (up to approximately 2.5 years)
  Adverse events during CDK4/6 regimen will be assessed according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided